CLINICAL TRIAL: NCT02305446
Title: Phase 3b, Open Label, Uncontrolled, Single-arm, Single-centre Study to Evaluate the Safety of Two Doses of Novartis Meningococcal Group B Vaccine When Administered to Healthy Adults From 18 to 50 Years of Age and to Collect Blood Donations to Develop Vaccines Against Neisseria Meningitidis
Brief Title: Safety and Blood Donations in Adults Vaccinated With rMenB+OMV NZ.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V72_74; 2014-002972-95 (EudraCT Number)
Record Dates: First submitted 2014-11-20; First posted 2014-12-02 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-12

CONDITIONS: Meningitis, Meningococcal, Serogroup B
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rMenB+OMV NZ (Experimental): Subjects who received two doses of rMenB+OMV NZ according to a 0, 2-month schedule
  Interventions: Biological: Meningococcal (group B) multicomponent recombinant adsorbed vaccine

INTERVENTIONS:
Biological: Meningococcal (group B) multicomponent recombinant adsorbed vaccine — One dose (0.5 mL) vaccine administered by intramuscular (IM) injection in the deltoid area of the non-dominant arm.
  Other Names: rMenB+OMV NZ

SUMMARY:
The purpose of this trial is to assess the safety of a Meningococcal Group B Vaccine and to collect blood donation. Sera panel obtained from blood donations will be used as a control to measure the immunoresponse to the Meningococcal Group B Vaccine in other studies.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals of 18 through 50 years of age on the day of informed consent;
2. Individuals who had voluntarily given written informed consent after the nature of the study had been explained according to local regulatory requirements, prior to study entry;
3. Individuals who could comply with study procedures including follow-up;
4. Males, females of non-childbearing potential or females of childbearing potential who are using an effective birth control method.

Exclusion Criteria:

1. Progressive, unstable or uncontrolled clinical conditions;
2. Hypersensitivity, including allergy, to any component of vaccines or medical equipment whose use is foreseen in this study;
3. Abnormal function of the immune system;
4. Chronic clinical significant conditions;

4. Been administered any group B meningococcal vaccine at any time prior to informed consent; 5. Current or previous, confirmed or suspected disease caused by N.meningitidis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- 01, Novartis Investigational Site, Krakow, Poland

REFERENCES:
- [Derived] Maritan M, Cozzi R, Lo Surdo P, Veggi D, Bottomley MJ, Malito E. Crystal structures of human Fabs targeting the Bexsero meningococcal vaccine antigen NHBA. Acta Crystallogr F Struct Biol Commun. 2017 Jun 1;73(Pt 6):305-314. doi: 10.1107/S2053230X17006021. Epub 2017 May 11. PMID 28580917

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be enrolled at one site in Poland from December 2014 to February 2015.
Pre-assignment Details: All enrolled subjects will be included in the trial and assigned to the same treatment group.
Period: Overall Study
Arm/Group | rMenB+OMV NZ
Started | 55
Completed | 54
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 27.2 (6.932)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs).
Description: Safety was assessed as the number of the subjects who reported unsolicited AEs following vaccination.
Time Frame: From day 1 to day 7 after each vaccination (Vaccination 1: Day 1 to Day 7; Vaccination 2: Day 61 to Day 67)
Population: Analysis were evaluated on the Unsolicited Safety Set
Measure: Number; unit: Subjects
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 55
Subjects
  Any Serious Adverse Events (SAEs) (vaccination 1) | 0
  Any Serious Adverse Events (SAEs) (vaccination 2) | 0
  At least possibly related SAEs (vaccination 1) | 0
  At least possibly related SAEs (vaccination 2) | 0
  AEs leading to premature withdrawal (vaccination1) | 0
  AEs leading to premature withdrawal (vaccination2) | 0
  Medically attended AEs (vaccination 1) | 0
  Medically attended AEs (vaccination 2) | 0
  AESIs (AEs of Special Interest) (vaccination 1) | 0
  AESIs (AEs of Special Interest) (vaccination 2) | 0

2. Other Pre Specified Outcome: Number of Adult Volunteers Whose Blood Can be Used as a Reference in Serum Bactericidal Activity (SBA) Test.
Description: The number of identified healthy adult volunteers with pre and postvaccination blood donations were summarized to establish a control sera panel to be used as a reference in SBA test.
Time Frame: Study day 1 blood sample was drawn between day -5 and day 1. Postvaccination 2 blood sample was drawn between day 23 and day 37 postvaccination 2.
Population: The analysis was performed on the all enrolled dataset.
Measure: Number; unit: Participants
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 55
Participants
  Study Day 1 Blood Sample | 55
  Postvaccination 2 Blood Sample | 50

ADVERSE EVENTS:
Time Frame: Safety was assessed from the day of first vaccination (Day 1) until and inclusive the day of study termination (pre-planned at Day 91).
Description: The analyses for unsolicited adverse events were done on the safety population. This study collects: throughout the study, any SAEs, AEs leading to withdrawal, AESI and medically attended AEs.
Arm/Group | rMenB+OMV NZ
Serious Adverse Events (participants affected / at risk) | 1/55
Other Adverse Events (participants affected / at risk) | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rMenB+OMV NZ (N=55)
MULTIPLE SCLEROSIS (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days